CLINICAL TRIAL: NCT06442722
Title: Evaluation of Surgical Treatment Outcomes for Developmental Dysplasia of Hip With and Without Capsulorrhaphy : a Comparative Study
Brief Title: Surgical Treatment of DDH With and Without Capsulorrhaphy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ali Abdelaal Bakheet, assistant lecturer, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Soh-Med-24-04-06MD
Record Dates: First submitted 2024-05-17; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Developmental Dysplasia of the Hip
MeSH Terms: conditions — Developmental Dysplasia of the Hip

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DDH with capsulorrhaphy (Active Comparator): one group will undergo capsulorrhaphy, a surgical procedure to tighten the hip capsule
  Interventions: Procedure: DDH with capsulorrhaphy
- DDH without capsulorrhaphy (Active Comparator): group has no tightness of the hip capsule
  Interventions: Procedure: DDH without capsulorrhaphy

INTERVENTIONS:
Procedure: DDH with capsulorrhaphy — group will undergo capsulorrhaphy, a surgical procedure to tighten the hip capsule ,
  Arms: DDH with capsulorrhaphy
Procedure: DDH without capsulorrhaphy — group will not undergo capsulorrhaphy, a surgical procedure without tightness the hip capsule
  Arms: DDH without capsulorrhaphy

SUMMARY:
The goal of this interventional study is to evaluates the surgical treatment outcomes of Developmental Dysplasia of Hip with and without capsulorrhaphy between 1-6 years of age . it compares the effectiveness of these approaches in improving postoperative stability , range of motion , and long-term success rates for DDH patients undergoing surgery .:

ELIGIBILITY:
Inclusion Criteria:

1. age: from 1 year to 6 years
2. sex: males and females
3. Children who received no operative treatment before.

Exclusion Criteria:

1. Children who were treated operatively before presentation.
2. Children who had teratologic, post septic or neuromuscular hip dislocation.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-06-02 (Estimated); Primary Completion 2025-06-02 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Severin's grading | 1 year
  radiological

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag Faculty Medicin, Sohag, Egypt